CLINICAL TRIAL: NCT00399360
Title: Strategies for the Treatment of HIV Associated Metabolic Syndrome
Brief Title: Lifestyle Modification and Metformin Use in the Treatment of HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK-49302-10AR; R01DK049302 (NIH)
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Metabolic Syndrome X
Keywords: HIV; Metabolic Syndrome; Lifestyle Modification; Metformin; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Placebo Comparator): No Lifestyle Modification and Placebo
  Interventions: Drug: Placebo
- Group 2 (Active Comparator): Lifestyle Modification and Placebo
  Interventions: Drug: Placebo; Behavioral: Lifestyle Modification
- Group 3 (Active Comparator): No Lifestyle Modification and Metformin
  Interventions: Drug: Metformin
- Group 4 (Active Comparator): Lifestyle Modification and Metformin
  Interventions: Drug: Metformin; Behavioral: Lifestyle Modification

INTERVENTIONS:
Drug: Metformin — Starting at 500 mg twice daily and increasing to 850 mg twice daily after 3 Months
  Arms: Group 3; Group 4
Drug: Placebo — 500 mg twice daily increasing to 850 mg twice daily after 3 Months
  Arms: Group 1; Group 2
Behavioral: Lifestyle Modification — Lifestyle Modification
  Arms: Group 2; Group 4

SUMMARY:
A healthy diet and exercise have improved the health of people without human immunodeficiency virus (HIV) who have Metabolic Syndrome. In this study we would like to find out if the same benefit can be seen in people with HIV and Metabolic Syndrome. Patients with Metabolic Syndrome usually have a large waist, high blood cholesterol levels, high blood pressure, and high blood sugar levels. These are risk factors, which may increase one's chance of developing heart disease and/or diabetes. The purpose of the study is to evaluate the effects of different methods of treating HIV associated Metabolic Syndrome. The groups are: 1) a lifestyle modification program plus metformin (also known as glucophage), 2) lifestyle modification plus placebo, 3) metformin alone or 4) placebo alone. The lifestyle modification program consists of nutrition and exercise sessions with the goal of improving body composition, heart health, and ways to lower the risk of developing diabetes.

DETAILED DESCRIPTION:
After two initial screening visits with medical and nutrition staff for informed consent and determination of eligibility qualifying subjects will be seen for a baseline visit.

At baseline subjects will have an interval history and physical exam, lipodystrophy evaluation by investigator and patient report. Bloods will be taken for insulin, glucose, HgbA1c, lipid studies, creatinine, liver function, serum lactate, urine pregnancy (women), CD4, viral load, and complete blood count (CBC). Metabolic assessment will include a 2-hour oral glucose tolerance test and indirect calorimetry. Carotid ultrasound will be done for assessment of intima-media thickness. Body composition will be assessed by dual energy x-ray absorptiometry (DEXA), single-slice magnetic resonance imaging (MRI) scanning through the abdomen and mid thigh, magnetic resonance spectroscopy scanning to assess intramyocellular lipid of the calf, anthropometric measurements, and Cardiac computed tomography (CT) will be done.

After the baseline visit, subjects will be randomized to 1 of 4 groups: 1) a lifestyle modification program plus metformin (also known as glucophage), 2) lifestyle modification plus placebo, 3) metformin alone or 4) placebo alone.

The starting dose of metformin will be 500mg twice daily and this will increase to 850mg twice daily at the 3-month visit.

An identical visit to that at baseline will be repeated at 12-months.

Subjects will return at 1 month for an interval history and physical exam, assessment of compliance and side effects. Blood will be collected for CBC, lactate, liver function, and creatinine. Women will have a urine pregnancy.

A 6-month visit will include an interval history and physical exam, assessment of compliance and side effects, 2 hour oral glucose tolerance test, fasting bloods (glucose, lipid panel, creatinine, liver function, serum lactate, CBC) will be done, a urine pregnancy will be checked in women. Carotid ultrasound will be done and body composition will be assessed by anthropometric measurements and DEXA scan.

There will also be a short visit at 3 and 9 months to obtain an interval history and physical exam, safety labs (serum lactate, CBC, liver function, and creatinine), urine pregnancy (women). Subjects randomized to metformin or placebo will increase their dose from 500mg twice daily to 850mg twice daily at the 3 month visit.

At each of the visits review of a 4 day food record will occur.

Those randomized to lifestyle modification will attend weekly sessions with a study investigator to cover a "core-curriculum" that is modeled after the Diabetes Prevention Program (DPP) intervention. The primary goals of the lifestyle modification program are derived from a combination of recommendations from the American Academy of Clinical Endocrinologists (AACE) and National Cholesterol Education Program (NCEP). The goals are to eat less than or equal to 35% of total calories from fat (less than 7% from saturated fat, up to 10% from polyunsaturated fat with emphasis on sources of omega 3 fatty acids and reduction of trans fatty acids, up to 20% from monounsaturated fats), and 25-35g of fiber per day.

The intensity of the counseling sessions will decrease in months 10 through 12 to biweekly counseling session with study investigators and biweekly phone contact, alternating.

In addition to the program outlined above, those randomized to the lifestyle modification group will also participate in progressive resistance training. Each training session will begin with a 5 minute warm-up on a stationary bicycle at 50% of the estimated maximal heart rate (maximal heart rate=220-age). All sessions will be monitored by a licensed physical therapist. Immediately after the warm-up, a standard flexibility routine will be performed to minimize the risk of injury. Then, the aerobic training protocol will be performed. The aerobic training program will follow the general guidelines established by the American College of Sports Medicine. Training will be performed using a standard stationary bicycle. Aerobic/endurance exercise will be performed with large muscle groups. Each subject will complete three supervised training sessions per week for 12 months.

Strength training will be performed using Keiser equipment. Selected muscle groups will be trained alternating upper and lower exercises in the following order: 1) hip extension, 2) lateral pull down, 3) knee extension, 4) elbow flexion, 5) knee flexion, and 6) chest press. Each repetition will include concentric and eccentric phases. Each muscle group will be trained individually 3 times per week, on alternate days. The subjects will perform three sets of 10 repetitions each for every muscle group, resting 2-3 seconds between repetitions, 2 minutes between sets, and 4 minutes between muscle groups. The 1 repetition maximum will be measured every 3-4 weeks for the first 6 months and it will be repeated again at the 9 and 12 month visits. The relative intensity will increase from 60-80% of the 1 repetition maximum over 6 months. Subjects not randomized to training will have a determination of 1 repetition maximum made at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65 years of age
* HIV positive, on a stable combination antiretroviral regimen for > 6 months, including but not limited to either 2 nucleoside reverse transcriptase inhibitors (NRTI) and a non-nucleoside reverse transcriptase inhibitors (NNRTI) or protease inhibitor (PI), or a triple NRTI regimen
* Ability and motivation to modify behavior and make lifestyle changes
* NCEP-Adult Treatment Panel III defined metabolic syndrome, as defined by 3 out of 5 of the following: 1) Waist circumference greater than 102 cm (40 in) in men and 88 cm (35 in) in women, 2) Triglycerides ≥ 150 mg/dL or current anti-lipolytic drug treatment, 3) high-density lipoprotein less than 40mg/dL in men and 50 mg/dL in women, 4) Blood pressure ≥ 130/85 mmHg or current antihypertensive drug treatment, 5) Fasting glucose ≥ 100 mg/dL

Exclusion Criteria:

* Any new serious opportunistic infection within the past 6 weeks
* History of unstable angina, aortic stenosis, uncontrolled hypertension, severe neuropathy, arthritis or other contraindication to exercise
* Current therapy with insulin or other diabetic agent, fasting blood sugar > 126
* Requiring parenteral nutrition or parenteral glucocorticoid therapy or oral glucocorticoid therapy
* Estrogen, progestational derivative, or ketoconazole use within 3 months
* New antiretroviral regimen in the past 6 months
* Serum creatinine > 1.5 mg/dL (males) and 1.4 mg/dL (females), serum glutamic pyruvic transaminase-liver function (SGPT), > 2.5 upper limit of normal (ULN), Lactate > 2.0 ULN, hemoglobin < 10.0 mg/dL
* Current substance and/or alcohol abuse
* Known hypersensitivity to Metformin
* Congestive heart failure requiring pharmacologic treatment
* Use of cimetidine or planned use during the study period
* Hypertrophic obstructive cardiomyopathy
* Pregnant or actively seeking pregnancy, breastfeeding
* Testosterone use for non-physiologic purposes, or physiologic testosterone replacement for < 3 months.
* Presence of active AIDS including cancers
* Current viral, bacterial or other infections (excluding HIV)
* Weight loss in the past 3 months of greater than 10 pounds
* Nitrates or other medications that can alter endothelial function
* Contraindication to beta blocker or nitroglycerin use
* Patients with previous allergic reactions to iodine-containing contrast media or to iodine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fitch K, Abbara S, Lee H, Stavrou E, Sacks R, Michel T, Hemphill L, Torriani M, Grinspoon S. Effects of lifestyle modification and metformin on atherosclerotic indices among HIV-infected patients with the metabolic syndrome. AIDS. 2012 Mar 13;26(5):587-97. doi: 10.1097/QAD.0b013e32834f33cc. PMID 22112605

RESULTS

PARTICIPANT FLOW:
Groups:
- No Lifestyle Modification and Placebo: Participants did not participate in lifestyle modification and took a placebo capsule 500mg twice daily x 3 months, which was increased to 850mg twice daily at the 3 month visit for the duration of the study.
- Lifestyle Modification and Placebo: Participants participated in lifestyle modification sessions 3 times a week for the duration of the study and took a placebo capsule 500mg twice daily for 3 months which was increased to 850mg twice daily at the 3 month visit for the duration of the study.
- No Lifestyle Modification and Metformin: Participants did not participate in lifestyle modification and took metformin 500mg twice daily for 3 months, this was increased to 850mg twice daily at the 3 month visit for the duration of the study.
- Lifestyle Modification and Metformin: Participants participated in lifestyle modification sessions 3 times a week for the duration of the study and took metformin 500mg twice daily for 3 months which was increased to 850mg twice daily at the 3 month visit for the duration of the study.
Period: Overall Study
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Started | 11 | 11 | 13 | 15
Completed | 9 | 8 | 10 | 9
Not Completed | 2 | 3 | 3 | 6
Not completed — Lost to Follow-up | 2 | 1 | 2 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin | Total
Number analyzed (Participants) | 11 | 11 | 13 | 15 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 13 | 15 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (6) | 49 (8) | 45 (9) | 47 (8) | 47 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 2 | 12
  Male | 7 | 8 | 10 | 13 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 5 | 16
  White | 7 | 6 | 9 | 10 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 13 | 15 | 50

OUTCOME MEASURES:

1. Primary Outcome: Carotid Intima Media Thickness
Description: Carotid intima media thickness imaging of the common carotid artery was conducted using a high-resolution 7.5-MHz phased-array transducer (SONOS 2000/2500. The change of the carotid intima media thickness measurement between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Population: All data were included in the analysis by intention to treat principle. For participants who did not complete a 12-month visit, last observation carried forward was performed for those participants for whom interim data post the baseline visit was available.
Measure: Mean (Standard Error); unit: mm
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
mm | -0.02 (0.03) | -0.02 (0.04) | 0.00 (0.01) | 0.03 (0.02)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.37, ANOVA

2. Primary Outcome: Waist Circumference
Description: Iliac waist circumference measurements were obtained using an inelastic tape measure. All measurements were obtained in triplicate, with the patient undressed, and then averaged. The change of the waist circumference measurement between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
cm | -1.9 (1.4) | -0.1 (1.7) | 0.3 (2.0) | -1.4 (1.8)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.80, ANOVA

3. Primary Outcome: High Density Lipoprotein (HDL)
Description: High density lipoprotein (HDL) was determined after an overnight fast. The change in HDL between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
mg/dL | -2 (1) | 2 (1) | 0 (2) | 4 (1)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.08, ANOVA

4. Primary Outcome: Glucose
Description: Glucose level was determined after an overnight fast. The change in glucose between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- No Lifestyle Modification and Placebo: All data were included in the analysis by intention to treat principle. For participants who did not complete a 12-month visit, last observation carried forward was performed for those participants for whom interim data post the baseline visit was available.
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
mg/dL | -7 (5) | 3 (3) | 2 (2) | -7 (3)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.13, ANOVA

5. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure was measured after 5 minutes rest. The in systolic blood pressure between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
mm Hg | -5 (4) | -2 (6) | -2 (4) | -6 (4)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.85, ANOVA

6. Primary Outcome: Coronary Artery Calcium Score
Description: Computed tomography (CT) imaging was performed using a SOMATOM Sensation (Siemens Medical Solutions, Forcheim, Germany) 64-slice CT scanner. Agatston calcium score was calculated using CT images. The total Agatston score is calculated by summing up the scores of the individual calcifications in all slices of the CT scan. An absolute Agatston score of less than 10 indicates minimal overall atherosclerosis (plaques) in the coronary arteries. The change in the coronary artery calcium score between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Agatston score
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
Agatston score | 43 (30) | 19 (7) | 1 (1) | -4 (6)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.03, ANOVA

7. Secondary Outcome: C-reactive Protein
Description: High sensitivity C-reactive protein was determined by R&D Systems (Minneapolis, MN) kit. The change in C-reactive protein between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Measure: Mean (Standard Error); unit: mg/l
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
mg/l | -0.27 (0.66) | -1.19 (1.11) | 0.47 (0.60) | -1.92 (0.93)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.10, ANOVA

8. Secondary Outcome: Abdominal Visceral Adiposity
Description: Abdominal visceral adipose area was assess by magnetic resonance imaging at the lvel of the L4 pedicle. The change in abdominal visceral adiposity between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Measure: Mean (Standard Error); unit: cm2
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
cm2 | -22.6 (14.5) | -1.5 (14.0) | -28.2 (15.3) | -35.0 (27.7)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.63, ANOVA

9. Secondary Outcome: Cardiorespiratory Fitness
Description: A submaximal exercise stress test was conducted on a cycle ergometer to measure endurance. Subjects cycled between 50-60 revolutions per minute and the workload was progressively increased in increments of 50 watts in stages lasting 3 minutes. Once subjects became fatigued or reached their submaximal heart rate (220-age x 85), the test was stopped and separate readings of heart rate and blood pressure were measured at 1, 3, and 5 min of recovery. Weight-adjusted maximum oxygen consumption (VO2max; ml/kg per minute) was determined. The change in cardiorespiratory fitness between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ml/kg/min
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
ml/kg/min | -0.7 (1.6) | 2.0 (1.2) | -1.3 (0.9) | 3.7 (1.8)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.05, ANOVA

10. Secondary Outcome: Intramyocellular Lipid
Description: Intramyocellular lipid (IMCL) of the tibialis anterior was determined using 1H-magnetic resonance spectroscopy (Siemens, Munich, Germany). The change in the intramyocellular lipid measurement between baseline and 12 months is reported.
Time Frame: baseline and 12 months
Measure: Mean (Standard Error); unit: mmol/kg
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Number analyzed (Participants) | 11 | 10 | 10 | 11
mmol/kg | 0.6 (0.2) | -0.4 (0.2) | 0.8 (0.4) | 0.1 (0.2)
Statistical Analysis 1: Comparison: No Lifestyle Modification and Placebo vs Lifestyle Modification and Placebo vs No Lifestyle Modification and Metformin vs Lifestyle Modification and Metformin; Test type: Superiority or Other; p = 0.02, ANOVA

ADVERSE EVENTS:
Time Frame: 12 months
Description: safety visits occurred at 1, 3, 6, and 9 months during which time ALT, creatinine, lactate level and CBC were checked
Arm/Group | No Lifestyle Modification and Placebo | Lifestyle Modification and Placebo | No Lifestyle Modification and Metformin | Lifestyle Modification and Metformin
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/11 | 2/11 | 3/13 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Lifestyle Modification and Placebo (N=11) | Lifestyle Modification and Placebo (N=11) | No Lifestyle Modification and Metformin (N=13) | Lifestyle Modification and Metformin (N=15)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
elevated creatinine (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was relatively small and may have been underpowered to assess effect on secondary endpoints and to assess the effects of lifestyle modification. The sample size may have limited our ability to determine differences in dropout rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No